CLINICAL TRIAL: NCT03120351
Title: Lidocaine 5% Patch (Lidoderm) for the Perioperative Prevention of Acute and Chronic Chest Pain Following Robotic Valve Surgery
Brief Title: Lidocaine 5% Patch (Lidoderm) for the Prevention of Acute and Chest Pain Following Robotic Valve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-379
Record Dates: First submitted 2017-03-21; First posted 2017-04-19 (Actual); Results first posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Perioperative Chest Pain
MeSH Terms: interventions — Lidoderm; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine patch 5% (Experimental): 1) Group I: Patients will receive topical 5% lidocaine patches. Those will be placed to affected area up to three patches as needed for pain 12 hours on and 12 hours off. They will also receive opioids as needed after the surgery. Initially, they may receive IV fentanyl repeated clinician boluses, later oxycodone will be given 5-10 mg q4-6 hours as needed for pain.
  Interventions: Drug: Lidoderm 5 % Topical Patch
- Placebo Patch (Placebo Comparator): 2) Group II: Patients will receive placebo patches. Those will be placed to affected area at dose up to three patches as needed for pain 12 hours on and 12 hours off. They will also receive opioids as needed after the surgery. Initially, they may receive IV fentanyl clinician boluses, later oxycodone will be given in doses from 5-10 mg q4-6 hours as needed for pain.
  Interventions: Drug: Placebo patch

INTERVENTIONS:
Drug: Lidoderm 5 % Topical Patch — Patients will receive Lidoderm topical 5% lidocaine patches. Those will be placed to affected area up to three patches as needed for pain 12 hours on and 12 hours off
  Other Names: Lidoderm
  Arms: Lidocaine patch 5%
Drug: Placebo patch — 2) Group II: Patients will receive placebo patches. Those will be placed to affected area at dose up to three patches as needed for pain 12 hours on and 12 hours off
  Arms: Placebo Patch

SUMMARY:
The post-thoracotomy pain (PTP) has been defined as persistent or recurrent pain that lasts for at least 2 month after thoracotomy and is associated with surgical incision or its intercostal nerve cutaneous distribution. The latter has a prevalence of about 15% to 20%. In about 80% of the patients such pain is moderate to severe in intensity and is associated with depression and insomnia. According to its characteristics and possible etiology, PTP is part of the neuropathic pain syndromes. Patients describe their chest wall pain as shooting, burning and numbness which are descriptors often seen in other neuropathic pain syndromes. PTP occurs most likely after partial or complete intercostal nerve damage secondary mechanical trauma (nerve traction or compression) during surgery. The concern is that when robotic surgery for minimally invasive approach to the heart valves or vessels such compression and consequent damage may happen to intercostal nerves.

Therapeutic use for a lidocaine patch include post-herpetic neuralgia postthoracotomy pain, stump neuroma pain, intercostal neuralgia, diabetic polyneuropathy, meralgia paresthetica, complex regional pain syndrome, radiculopathy, postmastectomy pain and some other focal peripheral neuropathic pain syndromes. It is an effective and safe topical treatment. Its efficacy demonstrated previously in treatment of intercostal neuralgia and some patients with post-thoracotomy syndrome can be used in treatment of perioperative chest pain related to robotic cardiac surgery. Hypothesis is that the use of topical lidocaine will decrease pain in acute phase after the surgery and decrease intensity of post-thoracotomy pain 6 months after such procedure.

The effect of topical 5% lidocaine will be clinically evaluated through prospective, randomized, placebo, double-blind study. Each patient will be assessed at admission and then, one week after Valve Replacement (Recommended surgical procedures do not included harvesting of leg vessels as this could be a potential confounder). Then, one month, three and six month follow-up for all patients by mailing questionnaires and phone calls.

Upon admission, as well as 1 week, 1month, 3months and 6 months following surgical procedure, the following tests will be performed:

* Pain Disability Index (PDI)
* DASS
* VAS Pain Score
* Opioid use (in MSO4 mg equivalents)
* Global Perceived Effect (GPE) or patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* consenting patients ≥ 18 years of age
* scheduled for robotic heart surgery

Exclusion Criteria:

Patient will be excluded from this study if they meet any of the following criteria:

* Patients with a history of mental instability or diagnosed with a mental disorder (e.g. Depression, Somatoform Conversion Disorder, Borderline Personality Disorder, etc.)
* Patients addicted to alcohol, narcotics and other illegal substances
* Patients with a known history of sensitivity to local anesthetics of the amide type, or to any other component of the product.
* Patients with severe hepatic disease (assessment by GI specialist)
* Pregnant Patients
* Patients less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 80 Enrolled
Period: Overall Study
Arm/Group | LIDOCAINE PATCH 5% | Placebo Patch
Started | 40 | 40
Completed | 39 | 39
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LIDOCAINE PATCH 5% | Placebo Patch | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (11) | 58 (10) | 57 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 31 | 29 | 60
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 26 (4) | 25 (4) | 26 (4)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 125 (16) | 126 (14) | 126 (15)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 72 (12) | 70 (10) | 71 (11)

OUTCOME MEASURES:

1. Primary Outcome: Pain Disability Index Score (PDI) at Six Months Following Surgical Procedure
Description: Pain Disability Index score (PDI) ranges from 0 to 70, with higher scores reflecting higher interference of pain with daily activities.
Time Frame: After surgery until postoperative day 7, 30, 90 and 180
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LIDOCAINE PATCH 5% | Placebo Patch
Number analyzed (Participants) | 39 | 39
units on a scale
  PDI on postoperative day 7 | 26 (17) | 30 (19)
  PDI on postoperative day 30 | 12 (14) | 13 (16)
  PDI on postoperative day 90 | 3.2 (7.8) | 5.0 (13.3)
  PDI on postoperative day 180 | 1.7 (6.4) | 4.8 (15.5)
Statistical Analysis 1: Comparison: LIDOCAINE PATCH 5% vs Placebo Patch; Test type: Superiority; p = 0.28, Mixed Models Analysis; Mean Difference (Net) = -2.5, 95% CI 2-sided [-7.11 to 2.06]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | LIDOCAINE PATCH 5% | Placebo Patch
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 3/39 | 2/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LIDOCAINE PATCH 5% (N=39) | Placebo Patch (N=39)
confusion (Nervous system disorders) | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LIDOCAINE PATCH 5% (N=39) | Placebo Patch (N=39)
Confusion (Nervous system disorders) | 1 | 0
atrial arrhythmia (Cardiac disorders) | 1 | 0
neurological deficit (Nervous system disorders) | 1 | 0
Ches wall hernia (General disorders) | 0 | 1
Pleural effusion (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Original PI (L. Kapural) and second PI (B. Vrooman) are no longer working at ClevelandCF

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes